CLINICAL TRIAL: NCT06760481
Title: Phase I/Ib Trial of TIraGolumab, AtEzolizumab, and RadScopal Radiation in Patients With Advanced Solid Malignancies (TIGER)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0309; NCI-2024-10794 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-12-31; First posted 2025-01-06 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Malignancies
MeSH Terms: interventions — Tiragolumab; atezolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- PhI/PhIbP1 Tiragolumab + Atezolizumab + RadScopal XRT (Experimental): Participants will be randomized to the trial using the Clinical Trial Conduct website
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Radiation: Radiation Therapy
- PhIbP2ArmA Atezolizumab + RadScopal XRT (Experimental): Participants will be randomized to the trial using the Clinical Trial Conduct website
  Interventions: Drug: Atezolizumab; Radiation: Radiation Therapy
- PhIbP2ArmB Tiragolumab + Atezolizumab + RadScopal XRT (Experimental): Participants will be randomized to the trial using the Clinical Trial Conduct website
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Radiation: Radiation Therapy
- PhIbP2ArmC Tiragolumab + Atezolizumab (Experimental): Participants will be randomized to the trial using the Clinical Trial Conduct website
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab

INTERVENTIONS:
Drug: Tiragolumab — Given by IV
  Arms: PhI/PhIbP1 Tiragolumab + Atezolizumab + RadScopal XRT; PhIbP2ArmB Tiragolumab + Atezolizumab + RadScopal XRT; PhIbP2ArmC Tiragolumab + Atezolizumab
Drug: Atezolizumab — Given by IV
Radiation: Radiation Therapy — Given by IV
  Arms: PhI/PhIbP1 Tiragolumab + Atezolizumab + RadScopal XRT; PhIbP2ArmA Atezolizumab + RadScopal XRT; PhIbP2ArmB Tiragolumab + Atezolizumab + RadScopal XRT

SUMMARY:
An open-label, Phase I/Ib study investigating the safety and efficacy of tiragolumab + atezolizumab + RadScopal™ XRT in patients with metastatic solid malignancies.

DETAILED DESCRIPTION:
Primary Objectives:

1. To evaluate the safety of tiragolumab + atezolizumab + RadScopal™ XRT (Phase I).
2. To evaluate the efficacy of tiragolumab + atezolizumab + RadScopal™ XRT (Phase Ib).

Secondary Objectives:

1. To compare the efficacy of tiragolumab + atezolizumab + RadScopal™ XRT to tiragolumab + atezolizumab and atezolizumab + RadScopal™ XRT.
2. To evaluate time-to-event outcomes of tiragolumab + atezolizumab + RadScopal™ XRT.

ELIGIBILITY:
Inclusion Criteria:

Aged ≥18 years at the time of informed consent form signing Patients must have a histologically confirmed metastatic or unresectable solid tumor.

1. All histological types will be eligible, with preference given to squamous histologies including lung, cervical, head and neck, and esophageal cancers.
2. Patients must not have available standard of care options or available standard of care option(s) are deemed to be less effective than the clinical trial alternative by the treating physician.
3. Life expectancy ≤3 months.
4. Prior anti-PD-1/PD-L1 therapy is allowed.
5. Patients will be eligible regardless of the number of prior lines of therapy.
6. Patients must have measurable disease per the RECIST v1.1.
7. Patients must have at least three active lesions, with at least one lesion amenable to HD-XRT (50 Gy in 4 fractions or 30 Gy in 5 fractions) as determined by the radiation oncologist. Repeat radiation with LD-XRT to previously irradiated sites will be allowed at the discretion of the investigator or treating radiation oncologist.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix A).
9. Adequate organ and marrow function as defined below:

Table 1. Adequate Organ Function Laboratory Values Systemic Function Test - Laboratory Value Hematologic ANC ≥1500/L Platelets ≥100,000/L Hemoglobin ≥9.0 g/dL Lymphocyte count ≥500/L Renal CrCl by Cockcroft-Gault formula

≥45 mL/min Hepatic Total bilirubin ≤1.5 × ULN (Patients with known Gilbert disease: ≤3 × ULN) AST, ALT, and ALP ≤2.5 × ULN (≤5 × ULN for patients with liver metastases) Albumin ≥2.5 g/dL Coagulation PT/INR aPTT ≤1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

aPTT=activated partial thromboplastin; ALP=alkaline phosphatase; ALT=alanine aminotransferase; ANC=absolute neutrophil count; AST=aspartate aminotransferase; CrCl=creatinine clearance; INR=international normalized ratio; PT=prothrombin time; ULN=upper limit of normal.

1. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen.
2. Negative hepatitis B surface antigen (HBsAg) test at screening. Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following:

   * Negative total hepatitis B core antibody (HBcAb).
   * Positive total HBcAb test followed by quantitative hepatitis B virus (HBV) DNA <500 IU/mL. NOTE: The HBV DNA test will be performed only for patients who have a negative HBsAg test, a negative HBsAb test, and a positive total HBcAb test.
3. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
4. Negative human immunodeficiency virus (HIV) test at screening with the following exception: individuals with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4+ T cell count ≥200/L, and have an undetectable viral load.
5. Patients with previously treated brain metastases may participate if they completed radiation therapy, are clinically stable, and without requirement of steroid treatment for at least 2 weeks prior to study enrollment.
6. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association (NYHA) Functional Classification. To be eligible for this trial, patients should have NYHA functional classification of 2B or better.
7. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test within 72 hours prior to study treatment initiation. If a WOCBP has a urine pregnancy test that cannot be confirmed as negative, a serum (beta-human chorionic gonadotropin [β-hCG]) pregnancy test will be required.
8. The effects of tiragolumab and atezolizumab on the developing human fetus are unknown. For this reason and because tiragolumab and atezolizumab as well as other therapeutic agents used in this trial are known to be teratogenic, WOCBP must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of the study treatment period, and for 90 days after the final dose of tiragolumab and 5 months after the final dose of atezolizumab. (Refer to Pregnancy Assessment Policy MDACC Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor, which may be one of the following:

<!-- -->

1. Postmenopausal (no menses in ≥12 consecutive months). History of hysterectomy or bilateral salpingo-oophorectomy.
2. Ovarian failure (follicle-stimulating hormone and estradiol in menopausal range and have received whole pelvic radiation therapy). History of bilateral tubal ligation or another surgical sterilization procedure.

   * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device, tubal ligation or hysterectomy, subject/partner post vasectomy, implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the study and the drug washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
   * Men must agree to remain abstinent (refrain from heterosexual intercourse) or use a condom plus spermicide, and agree to refrain from donating sperm, as defined below:

   With a female partner of childbearing potential, men who are not surgically sterile must remain abstinent or use a condom plus spermicideduring the study treatment period and for 90 days after the final dose of tiragolumab. Men mustrefrain from donating sperm during this same period.

   With a pregnant female partner, men must remain abstinent or use a condom plus spermicide during the treatment period for 90 days after the final dose of tiragolumab.
   * Ability to understand and the willingness to sign a written informed consent document.
   * Ability to comply with the study protocol.

   Exclusion Criteria:

   History of leptomeningeal disease. ● Uncontrolled tumor-related pain Patients requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.

   Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
   * Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX®) are allowed.
   * Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmo1/L, calcium >12 mg/dL or corrected serum calcium > ULN).
   * Active tuberculosis.
   * Received XRT within 14 days prior to study treatment initiation.
   * Received anticancer systemic therapies (including chemotherapy, immunotherapy, targeted therapy, or other modalities such as investigational agents) within 21 days or 5 half-lives of the drug, whichever is shorter.
   * Prior XRT to the target lesion(s) selected for HD-XRT. Previous radiation to LDXRT target lesions is allowed per investigator or treating radiation oncologist discretion.
   * Unresolved Grade ≥2 AEs from prior anticancer therapy. Patients with Grade 2 neuropathy, alopecia, or other non-relevant AEs may be deemed eligible at the discretion of the principal investigator (PI).
   * Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or tiragolumab formulation.
   * History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
   * Requirement for systemic IV antibiotics for infection within 3 days prior to study treatment initiation. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
   * Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment, within 90 days after the final dose of tiragolumab, or within 5 months after the final dose of atezolizumab.
   * Positive Epstein-Barr virus (EBV) viral capsid antigen IgM test at screening. An EBV polymerase chain reaction (PCR) test should be performed as clinically indicated to screen for acute infection or suspected chronic active infection. Patients with a positive EBV PCR test are excluded.
   * Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, renal failure, cardiac arrhythmia, or psychiatric illness that would adversely impact the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures, or interpretation of study results.
   * History of severe (Grade ≥3) imAEs observed with previous PD-1/L1 ICI that led to treatment discontinuation and rechallenge with ICI was not possible.
   * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
   * Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (see Appendix C for a more comprehensive list of autoimmune diseases and immune deficiencies), with the exceptions listed below:
   * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
   * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   * Patients with eczema, psoriasis lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met: - Rash must cover <10% of body surface area.

     - Disease is well controlled at baseline and requires only low-potency topical corticosteroids.

   There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.

   ● Significant cardiovascular disease (such as NYHA Class 2 or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.

   ● Major surgical procedure within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study.

   ● History of malignancy within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.

   ● Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety.

   ● Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
   * Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin-2) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to study treatment initiation.
   * Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to study treatment initiation, with the following exceptions:

     * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
     * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or lowdose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
   * Prior allogenic stem cell transplantation or organ allograft.
   * Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment and within 90 days after the final dose of tiragolumab and 5 months after the final dose of atezolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2025-04-13 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2030-09-15 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ecaterina Dumbrava, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org